CLINICAL TRIAL: NCT03948334
Title: A Randomized, Double Blind, Multicenter Extension to CZPL389A2203 Dose-ranging Study to Assess the Short-term and Long-term Safety and Efficacy of Oral ZPL389 With Concomitant Use of TCS and/or TCI in Adult Patients With Atopic Dermatitis.
Brief Title: A Study to Assess the Safety and Efficacy of ZPL389 With TCS/TCI in Atopic Dermatitis Patients
Acronym: ZESTExt
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Core terminated due to lack of efficacy
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZPL389A2203E1; 2018-000595-15 (EudraCT Number)
Record Dates: First submitted 2019-04-04; First posted 2019-05-13 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; AD; eczema; itch; pruritus; H4R; ZPL389
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZPL389 30mg (Experimental): 30mg of ZPL389 + TCS and/or TCI for patients re-randomized from the core study (received placebo/ZPL389 3mg/ 10mg in the core study) and for patients continuing in the same arm from the core study
  Interventions: Drug: ZPL389 30mg; Drug: TCS and/or TCI
- ZPL389 50mg (Experimental): 50mg of ZPL389 + TCS and/or TCI for patients re-randomized from the core study (received placebo/ZPL389 3mg/ 10mg in the core study) and for patients continuing in the same arm from the core study
  Interventions: Drug: ZPL389 50mg; Drug: TCS and/or TCI

INTERVENTIONS:
Drug: ZPL389 30mg — 30mg of ZPL389; once daily
  Arms: ZPL389 30mg
Drug: ZPL389 50mg — 50mg of ZPL389; once daily
  Arms: ZPL389 50mg
Drug: TCS and/or TCI — Topical corticosteroids (TCS) and /or topical calcineurin inhibitors (TCI) were used concomitantly or intermittently based on disease severity.

SUMMARY:
This extension study (CZPL389A2203E1) was designed as a 2-year (100 weeks) extension to the core study (CZPL389A2203/ NCT03517566) which is disclosed separately. It aimed to assess the short-term and long-term safety of (blinded) 30 mg o.d and 50 mg o.d ZPL389 with concomitant or intermittent use of topical corticosteroids (TCS) and/or topical calcineurin inhibitors (TCI).

DETAILED DESCRIPTION:
Subjects who had received ZPL389 30 mg or 50 mg doses in the core study (CZPL389A2203), continued to receive the same doses in double-blinded fashion. Subjects who had received ZPL389 3 mg, 10 mg or placebo in the core study were randomized to 30 mg or 50 mg ZPL389 in a 1:1 ratio. All subjects received concomitant or intermittent TCS and/or TCI along with ZPL389. Short-term safety was assessed up to week 16 of this extension study (week 16 to week 32 referring to the start of core study treatment) and long-term safety was assessed after week 16 of this extension study (after week 32 referring to the start of core study treatment). The entire planned time frame (100 weeks) was not assessed as originally planned due to early termination of the core and extension studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give a written, signed and dated informed consent
* Subjects with atopic dermatitis who have participated in and completed 16 weeks of treatment in CZPL389A2203 study.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, diary completion and other study procedures.

Exclusion Criteria:

* Inability to use TCS and/or TCI due to history of important side effects of topical medication (e.g., intolerance or hypersensitivity reactions).
* Treatment discontinued subject from CZPL389A2203 study.
* Any skin disease that would confound the diagnosis or evaluation of atopic dermatitis disease activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (2):
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Fairborn, Ohio
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Turku
- Germany (9):
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
- Novartis Investigative Site, Kopavogur, Iceland
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Bergen op Zoom
- Poland (3):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (5):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
- Slovakia (4):
  - Novartis Investigative Site, Bardejov, SVK
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Svidník
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=725

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who had received ZPL389 30 mg or 50 mg doses in the core study, continued to receive the same doses in double-blinded fashion.
  Subjects who had received ZPL389 3 mg, 10 mg or placebo in the core study were randomized to 30 mg or 50 mg ZPL389 in a 1:1 ratio.
Groups:
- ZPL389 30mg: Dose 1 of ZPL389 + TCS and/or TCI
- ZPL389 50mg: Dose 2 of ZPL389 + TCS and/or TCI
Period: Overall Study
Arm/Group | ZPL389 30mg | ZPL389 50mg
Started | 60 | 63
Completed | 0 | 0
Not Completed | 60 | 63
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Study terminated by Sponsor | 50 | 51
Not completed — Subject Decision /Guardian Decision | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZPL389 30mg | ZPL389 50mg | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.18) | 34.4 (11.24) | 34.6 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 36 | 43 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 42 | 78
  Black or African American | 1 | 1 | 2
  Asian | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events in the First 16 Weeks of This Extension Study
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study until the end of study visit. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  As all patients were rolling over from the core study CZPL389A2203, in addition to the time frame referring to the start in this extension study, the time frame corresponding to the start in the core study (+16 weeks) are provided in parenthesis.
Time Frame: 16 weeks (week 16 to week 32 referring to core study)
Population: The Extension study set comprised all subjects who were randomized and to whom study treatment had been assigned and had at least one visit in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 60 | 63
Participants
  Adverse events | 29 | 33
  SAEs | 2 | 5
  AEs leading to discontinuation | 2 | 3

2. Primary Outcome: Number of Patients With Adverse Events After 16 Weeks of Treatment in This Extension Study
Description: as for outcome 1
Time Frame: From week 16 to week 67 of this extension study (week 32 to week 83 referring to core study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- ZPL389 30mg: 30mg of ZPL389 + TCS and/or TCI
- ZPL389 50mg: 50mg of ZPL389 + TCS and/or TCI
Arm/Group | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 60 | 63
Participants
  Adverse events | 18 | 20
  SAEs | 0 | 2
  AEs leading to discontinuation | 0 | 1

3. Secondary Outcome: Percentage of Investigator's Global Assessment (IGA) Responders Over Time
Description: IGA score is used to determine the severity of atopic dermatitis symptoms and clinical response to treatment. The scale ranges from 0=clear to 4=severe. It is a static scale and doesn't refer to previous status of the subject. IGA response is an achievement of an IGA score of 0 or 1 with a 2-point reduction from baseline without use of confounding therapy up to the assessment time point. Treatment discontinuations for lack of efficacy or AE are considered non-responders.Presentation of the results is stratified by if patients were re-randomized from the core study or not. As all patients were rolling over from the core study, in addition to the timeframe referring to the start in this extension study, the timeframe corresponding to the start in the core study (+16 weeks) are provided in parenthesis. Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline IGA as covariates.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28, Week 40 (Week 20, Week 24, Week 28 ,Week 32, Week 44, Week 56 referring to core study)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- ZPL389 30mg Re-randomized After Core Study: 30mg of ZPL389 + TCS and/or TCI for patients re-randomized from the core study (received placebo/ ZPL389 3mg/ 10mg in the core study)
- ZPL389 50mg Re-randomized After Core Study: 50mg of ZPL389 + TCS and/or TCI for patients re-randomized from the core study (received placebo/ ZPL389 3mg/ 10mg in the core study)
- ZPL389 30mg Continuing After Core Study: 30mg of ZPL389 + TCS and/or TCI for patients continuing in the same arm from the core study
- ZPL389 50mg Continuing After Core Study: 50mg of ZPL389 + TCS and/or TCI for patients continuing in the same arm from the core study
Arm/Group | ZPL389 30mg Re-randomized After Core Study | ZPL389 50mg Re-randomized After Core Study | ZPL389 30mg Continuing After Core Study | ZPL389 50mg Continuing After Core Study
Number analyzed (Participants) | 34 | 30 | 26 | 33
Percentage of participants
  week 4 (week 20 referring to core study) | 2.9 [-2.7 to 8.6] | 5.2 [-3.4 to 13.8] | 0.0 [-0.0 to 0.0] | 3.0 [-2.8 to 8.9]
  Week 8 (week 24 referring to core study) | 2.9 [-2.7 to 8.6] | 4.8 [-3.9 to 13.5] | 0.0 [-0.0 to 0.0] | 3.1 [-2.8 to 9.0]
  Week 12 (week 28 referring to core study) | 3.5 [-3.1 to 10.1] | 4.0 [-4.4 to 12.4] | 0.0 [-1.0 to 1.1] | 3.0 [-2.8 to 8.9]
  Week 16 (week 32 referring to core study) | 3.9 [-3.3 to 11.0] | 5.9 [-3.7 to 15.5] | 0.0 [-1.7 to 1.9] | 0.0 [-2.0 to 2.4]
  Week 28 (week 44 referring to core study) | 0.0 [-3.7 to 6.4] | 7.5 [-3.7 to 18.7] | 0.0 [-1.4 to 1.6] | 1.5 [-3.8 to 6.9]
  Week 40 (week 56 referring to core study) | 3.4 [-4.4 to 11.2] | 9.1 [-2.7 to 20.8] | 0.0 [-4.3 to 7.0] | 0.0 [-4.2 to 7.0]

4. Secondary Outcome: Percentage of EASI50 Responders Over Time
Description: Eczema Area and Severity Index (EASI) is used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
  EASI50 response is defined as achieving ≥ 50% improvement (reduction) in EASI score compared to baseline.
  Treatment discontinuations for lack of efficacy or adverse event are considered non-responders.
  Presentation of the results is stratified by if patients were re-randomized from the core study or not.
  As all patients were rolling over from the core study CZPL389A2203, in addition to the time frame referring to the start in this extension study, the time frame corresponding to the start in the core study (+16 weeks) are provided in parenthesis.
  Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline EASI as covariates.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ZPL389 30mg Re-randomized After Core Study | ZPL389 50mg Re-randomized After Core Study | ZPL389 30mg Continuing After Core Study | ZPL389 50mg Continuing After Core Study
Number analyzed (Participants) | 34 | 30 | 26 | 33
Percentage of participants
  week 4 (week 20 referring to core study) | 14.7 [2.8 to 26.6] | 13.0 [0.8 to 25.2] | 7.7 [-2.6 to 17.9] | 12.1 [1.0 to 23.3]
  Week 8 (week 24 referring to core study) | 17.6 [4.8 to 30.5] | 15.6 [2.2 to 29.0] | 11.5 [-0.7 to 23.8] | 12.1 [1.0 to 23.3]
  Week 12 (week 28 referring to core study) | 22.3 [8.0 to 36.6] | 15.9 [2.5 to 29.3] | 10.7 [-1.5 to 23.0] | 12.1 [1.0 to 23.3]
  Week 16 (week 32 referring to core study) | 19.6 [5.7 to 33.4] | 18.2 [3.8 to 32.6] | 10.1 [-2.0 to 22.2] | 11.9 [0.5 to 23.3]
  Week 28 (week 44 referring to core study) | 10.8 [-1.0 to 22.6] | 14.8 [0.8 to 28.8] | 14.0 [0.1 to 27.8] | 14.2 [1.6 to 26.8]
  Week 40 (week 56 referring to core study) | 14.8 [1.4 to 28.2] | 20.3 [4.6 to 36.1] | 12.3 [-0.9 to 25.5] | 13.8 [0.9 to 26.6]

5. Secondary Outcome: Percentage of EASI75 Responders Over Time
Description: Eczema Area and Severity Index (EASI) is used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
  EASI75 response is defined as a reduction from baseline of ≥ 75% in EASI score. Treatment discontinuations for lack of efficacy or adverse event are considered non-responders.
  Presentation of the results is stratified by if patients were re-randomized from the core study or not.
  As all patients were rolling over from the core study CZPL389A2203, in addition to the time frame referring to the start in this extension study, the time frame corresponding to the start in the core study (+16 weeks) are provided in parenthesis.
  Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline EASI as covariates.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ZPL389 30mg Re-randomized After Core Study | ZPL389 50mg Re-randomized After Core Study | ZPL389 30mg Continuing After Core Study | ZPL389 50mg Continuing After Core Study
Number analyzed (Participants) | 34 | 30 | 26 | 33
Percentage of participants
  week 4 (week 20 referring to core study) | 5.9 [-2.0 to 13.8] | 8.8 [-1.8 to 19.4] | 0.0 [-0.0 to 0.0] | 12.1 [1.0 to 23.3]
  Week 8 (week 24 referring to core study) | 5.9 [-2.0 to 13.8] | 14.2 [1.0 to 27.4] | 0.0 [-0.0 to 0.0] | 9.1 [-0.7 to 18.9]
  Week 12 (week 28 referring to core study) | 12.0 [1.0 to 23.1] | 11.4 [-0.6 to 23.4] | 4.6 [-4.0 to 13.2] | 12.1 [1.0 to 23.3]
  Week 16 (week 32 referring to core study) | 8.4 [-1.8 to 18.7] | 10.3 [-1.3 to 22.0] | 0.0 [-4.2 to 6.6] | 4.9 [-3.0 to 12.8]
  Week 28 (week 44 referring to core study) | 8.2 [-2.0 to 18.5] | 8.9 [-2.9 to 20.8] | 0.0 [-4.0 to 5.9] | 2.6 [-4.6 to 9.9]
  Week 40 (week 56 referring to core study) | 10.0 [-2.4 to 22.3] | 13.5 [-0.2 to 27.3] | 6.1 [-4.0 to 16.2] | 3.2 [-4.4 to 10.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment in this extension study until end of study treatment plus 4 weeks post treatment, up to maximum duration of 67 weeks (week 16 to week 83 referring to core study).
Description: Any sign or symptom that occurs during the study treatment plus the 4 weeks post treatment
Groups:
- ZPL389 30mg in the First 16 Weeks of This Extension Study; ZPL389 50mg in the First 16 Weeks of This Extension Study: AEs starting up to week 16 of this extension study (week 16 to week 32 referring to core study)
- ZPL389 30 mg After 16 Weeks of Treatment in This Extension Study; ZPL389 50 mg After 16 Weeks of Treatment in This Extension Study: AEs from week 16 to week 67 of this extension study (week 32 to week 83 referring to core study)
Arm/Group | ZPL389 30mg in the First 16 Weeks of This Extension Study | ZPL389 50mg in the First 16 Weeks of This Extension Study | ZPL389 30 mg After 16 Weeks of Treatment in This Extension Study | ZPL389 50 mg After 16 Weeks of Treatment in This Extension Study
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/63 | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/60 | 5/63 | 0/60 | 2/63
Other Adverse Events (participants affected / at risk) | 6/60 | 8/63 | 9/60 | 6/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL389 30mg in the First 16 Weeks of This Extension Study (N=60) | ZPL389 50mg in the First 16 Weeks of This Extension Study (N=63) | ZPL389 30 mg After 16 Weeks of Treatment in This Extension Study (N=60) | ZPL389 50 mg After 16 Weeks of Treatment in This Extension Study (N=63)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL389 30mg in the First 16 Weeks of This Extension Study (N=60) | ZPL389 50mg in the First 16 Weeks of This Extension Study (N=63) | ZPL389 30 mg After 16 Weeks of Treatment in This Extension Study (N=60) | ZPL389 50 mg After 16 Weeks of Treatment in This Extension Study (N=63)
Nasopharyngitis (Infections and infestations) | 6 | 4 | 8 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03948334/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT03948334/SAP_001.pdf